CLINICAL TRIAL: NCT03570996
Title: A Randomized Controlled Trial Comparing Transversus Abdominis Plane Catheter Versus Epidural After Esophagectomy
Brief Title: A Trial Comparing Transversus Abdominis Plane Catheter Versus Epidural After Esophagectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID 19
Sponsor: Swedish Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY2017000592
Record Dates: First submitted 2018-03-21; First posted 2018-06-27 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Esophageal Cancer; Pain, Postoperative
Keywords: esophageal cancer; transversus abdominis plane catheter; epidural; pain, postoperative
MeSH Terms: conditions — Esophageal Neoplasms; Pain, Postoperative | interventions — Esophagectomy; Injections, Epidural; tetraethylpyrazine

STUDY DESIGN:
Intervention Model Description: Randomization into either transversus abdominis plane catheter (TAP) or epidural for patients undergoing esophagectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversus abdominis plane catheter (Active Comparator): Transversus abdominis plane catheter (TAP) for pain control in esophagectomy operations. TAP group will have bilateral subcostal TAP catheters and single shot bilateral rectus sheath blocks placed at the end of the surgery, prior to emergence. Bilateral subcostal TAP catheters will be bolused with 20ml of .2% ropivacaine on each side and then infused with .2% ropivacaine at 10ml/ hr for 75 hours each. Rectus sheath blocks will be bilateral bolus 20ml of .2% ropivacaine.
  Interventions: Procedure: Esophagectomy; Procedure: Transversus abdominis plane catheter
- epidural (Active Comparator): Epidural pain control for pain control in esophagectomy operation. Patients randomize the TEP group will have bilateral TEP placed at T8-9 +/- one level based on patient anatomy. TEP will be bolused with 5ml of 1.5% lidocaine with epinephrine and then started on infusion of .0625% bupivacaine plus 4 mcg/ml fentanyl plus 2 mcg/ ml epinephrine at 6ml/hr with a range of 6-12 ml/hr, titrating to optimize patient comfort. Epidurals are placed before surgery start time.
  Interventions: Procedure: Esophagectomy; Procedure: Epidural

INTERVENTIONS:
Procedure: Esophagectomy — Esophagectomy with minimally invasive approach of the chest including:
  3 hole with R video-assisted thoracoscopic surgery (VATS), Ivor Lewis R VATS, Transhiatal
Procedure: Transversus abdominis plane catheter — TAP group will have bilateral subcostal TAP catheters and single shot bilateral rectus sheath blocks placed at the end of the surgery, prior to emergence. Bilateral subcostal TAP catheters will be bolused with 20ml of .2% ropivacaine on each side and then infused with .2% ropivacaine at 10ml/ hr for 75 hours each. Rectus sheath blocks will be bilateral bolus 20ml of .2% ropivacaine
  Other Names: TAP catheter
  Arms: Transversus abdominis plane catheter
Procedure: Epidural — Patients randomize the TEP group will have bilateral TEP placed at T8-9 +/- one level based on patient anatomy. TEP will be bolused with 5ml of 1.5% lidocaine with epinephrine and then started on infusion of .0625% bupivacaine plus 4 mcg/ml fentanyl plus 2 mcg/ ml epinephrine at 6ml/hr with a range of 6-12 ml/hr, titrating to optimize patient comfort. Epidurals are placed before surgery start time.
  Other Names: TEP
  Arms: epidural

SUMMARY:
A randomized trial comparing perioperative outcomes between bilateral transversus abdominis plane TAP catheters with patient controlled analgesia (PCA) to epidural for esophagectomy patients with a VATS chest approach. Further objectives are to determine pain requirements between multiple modalities of pain control and compare the subsequent sequelae of narcotic use and blood pressure control and to compare complications such as anastomotic leak, atrial fibrillation and perioperative morbidity and mortality between the two groups.

DETAILED DESCRIPTION:
Epidural analgesia is considered the 'gold standard' for post-operative analgesia following open esophagectomy. Epidurals have been shown to reduce post-operative pulmonary morbidity and mortality. However, epidurals are often associated with sympathetic blockade that creates hypotension and could therefore adversely affect the conduit. Pain management techniques that use peripheral nerve blockade are becoming more prevalent, reducing the need for an epidural. Transversus abdominis plane (TAP) catheters have been used in colorectal and abdominal surgery showing equivocal pain scores to epidurals. With the minimally invasive chest approach, the analgesia coverage focuses on the abdominal incision where both epidurals and TAPs are considered standard of care.

The investigators have completed a retrospective study in preparation for a randomized control trial. The investigators previous retrospective study found that TAP blocks/catheters are a reasonable alternative to epidurals, providing adequate pain coverage for abdominal incisions. The study found no statistical difference in pain scores between the two groups. The TAP group had a lower prevalence of hypotension and lower crystalloid resuscitation needs. Pulmonary complications were similar between the two groups. This retrospective review showed that TAP blocks are a reasonable alternative to epidurals and may reduce episodes of hypotension. The investigators aim is to now expand this study to a randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

* All adult individuals who undergo an esophagectomy with a minimally invasive approach of the chest at Swedish Medical Center-First Hill. These approaches include:
* 3 hole with R video-assisted thoracoscopic surgery (VATS)
* Ivor Lewis R VATS
* Transhiatal

Exclusion Criteria:

* Age <18
* Unable to consent
* Additional surgical procedures planned
* Patient with chronic pain on a daily regimen of narcotics
* Patients who remain intubated greater than 24 hours post operatively
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Pain scores | Up to post-operative day 4
  Pain scores on a scale of 0-10 will be collected from patients twice a day

SECONDARY OUTCOMES:
Volume Resuscitation | Up to post-operative day 4
  Amount of fluids given to patient
Hypotension | Up to post-operative day 4
  Total episodes of hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Brian E Louie, MD, Principal Investigator — Swedish Cancer Institute and Medical Center
Locations (1):
- Swedish Cancer Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No